CLINICAL TRIAL: NCT06970158
Title: Effect of Automated AI Designed Presurgical Plate Therapy on Cleft Size Reduction in Newborns With Cleft Lip and Palate : A Comparative Study
Brief Title: Clinical Application of Artificial Intelligence in New Borns With Cleft Lip and Palate
Acronym: CLIP-AI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Principal Investigator, Prasad Nalabothu, Prinicipal Investigator, University Hospital, Basel, Switzerland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: placeholder unique ID
Record Dates: First submitted 2024-05-07; First posted 2025-05-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Congenital Disorder; Cleft Lip Palate
Keywords: artificial intelligence; Cleft Lip Palate
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups based on clinical site practices. The treatment group will receive AI-designed passive plate therapy from shortly after birth until primary surgery and will undergo intraoral scans at birth and at approximately 4 months of age. The comparison group will receive no presurgical intervention and will undergo a single intraoral scan at the time of primary surgery (around 4 months). This parallel design allows for evaluation of cleft size at surgery between treated and untreated groups.
Masking Description: No masking is implemented in this study. All parties, including care providers and outcome assessors, are aware of group assignments due to the nature of the intervention and clinical workflow.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Designed Passive Plate Therapy (Experimental): Infants in this group will receive passive plate therapy designed using an AI-assisted digital workflow. The plate is fitted shortly after birth and worn continuously until the time of primary surgical repair (around 4 months of age). Participants in this arm will undergo intraoral scans at birth and again at surgery.
  Interventions: Other: AI-Designed Passive Plate Therapy
- No Presurgical Therapy (No Intervention): Infants in this group will not receive any presurgical orthopedic intervention. They will undergo a single intraoral scan at the time of primary surgical repair (around 4 months of age), which will be used for comparison with the intervention group.

INTERVENTIONS:
Other: AI-Designed Passive Plate Therapy — A removable passive orthopedic plate designed using an AI-assisted digital workflow based on intraoral scan data. The design process is automated via a Blender-based software plugin that identifies anatomical landmarks and generates a custom-fit plate. The plate is 3D printed using biocompatible material and fitted shortly after birth. It is worn continuously until primary surgical repair, typically around 4 months of age. The intervention aims to reduce cleft width prior to surgery without requiring traditional impressions or extensive manual design effort.
  Other Names: Automated Passive Plate
  Arms: AI-Designed Passive Plate Therapy

SUMMARY:
The goal of this observational study is to evaluate whether passive plate therapy using automated AI-designed devices can reduce cleft size in newborns with cleft lip and palate. The main questions it aims to answer are:

Does AI-designed passive plate therapy reduce the cleft size between birth and primary surgery? (Primary aim)

How does cleft size at the time of surgery compare between infants who received passive plate therapy and those who did not? (Secondary aim)

Researchers will compare infants who received AI-designed passive plate therapy with those who received no presurgical therapy to determine whether the intervention leads to a greater reduction in cleft width.

Participants will: Undergo intraoral scans at birth and again at the time of primary surgery, around 4 months of age.

Receive either no presurgical intervention or be treated with AI-designed passive plates, depending on site-specific clinical practices

DETAILED DESCRIPTION:
This observational study investigates the impact of passive plate therapy using an automated, artificial intelligence (AI)-driven design workflow on presurgical cleft size in infants with unilateral cleft lip and palate. Cleft lip and palate represent one of the most common congenital craniofacial anomalies, and early presurgical interventions such as passive plates aim to reduce the cleft size, support feeding, and facilitate better surgical outcomes. However, access to such interventions is often limited by the need for specialized staff, complex workflows, and reliance on intraoral impressions.

Recent technological advancements have enabled the integration of digital workflows and AI into presurgical cleft care. In particular, a pipeline has been developed that uses intraoral scanning, and AI-assisted modeling to design individualized passive plates. These plates are manufactured via 3D printing and do not require invasive impressions nor extensive laboratory work making them potentially safer and more scalable in low or medium resource settings.

This study specifically evaluates the clinical effectiveness of such AI-designed passive plates compared to standard care without any presurgical orthopedic therapy. Infants are enrolled from two sites in India (Chennai and Hyderabad), where clinical practices differ with respect to the use of passive plates. As this is a non-randomized, observational study, group assignment is based on local standard of care at each site.

The primary objective is to assess the percentage reduction in cleft width from birth to the time of primary surgery (typically around 4 months of age) in infants treated with AI-designed passive plates. The secondary objective is to compare cleft width at the time of surgery between infants who received the plates and those who did not, offering insight into the relative anatomical outcomes of the intervention.

All participating infants will undergo standardized intraoral scans at baseline (within the first two weeks of life) and again just prior to primary surgical repair. The scans are used to measure the anterior-posterior cleft width and calculate percentage change over time. Cleft measurements are obtained digitally from 3D scan data using validated image processing software.

The AI-assisted design of the passive plates is performed using a custom plugin within Blender software, which automatically detects anatomical landmarks and generates the plate geometry with minimal user input. The digital files are subsequently exported for 3D printing using biocompatible materials. Infants in the intervention group will wear the plate continuously from the time of fitting until primary surgery, under the supervision of trained clinical teams.

Data from the two cohorts (plate vs. no plate) will be compared using appropriate statistical methods to assess differences in cleft size reduction and absolute cleft width at surgery. This study does not include randomization or blinding, as the intervention is assigned based on institutional practice. However, efforts will be made to ensure consistency in scanning methods, measurement protocols, and outcome assessment across both sites.

This study is part of a larger initiative to evaluate the generalizability and effectiveness of AI-based digital workflows in cleft care across diverse healthcare settings. The findings are expected to inform future integration of automated design technologies in presurgical treatment planning, especially in regions where access to skilled cleft teams is limited.

No additional interventions, medications, or behavioral changes are introduced as part of this study. Participation involves routine procedures and follow-up through the standard cleft treatment timeline.

ELIGIBILITY:
Inclusion criteria:

Infants diagnosed with unilateral cleft lip and palate Age at enrollment: within the first 14 days of life (for treatment group) Age at cleft surgery: approximately 4 months Medically stable and fit to undergo intraoral scanning and cleft surgery Parent or legal guardian has provided written informed consent

Exclusion Criteria:

Syndromic cleft lip and palate or other craniofacial syndromes Bilateral cleft lip and palate Significant comorbidities affecting feeding, growth, or surgery (e.g., cardiac anomalies) Premature infants (<37 weeks gestational age at birth) Infants who have already undergone any presurgical orthopedic intervention elsewhere Guardians/ Parents unwilling or unable to comply with follow-up or study procedures

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Reduction in Cleft Width from Birth to Primary Surgery | From birth to time of primary cleft surgery (approximately 4 months of age)
  Measured as the percentage change in anterior-posterior cleft width between the intraoral scan at birth and the scan at the time of primary surgery (~4 months), in infants receiving AI-designed passive plate therapy.

SECONDARY OUTCOMES:
Cleft Width at Time of Primary Surgery | At the time of primary cleft surgery (approximately 4 months of age)
  Absolute cleft width (in mm) at the time of primary surgery, measured from intraoral scan data. This will be compared between infants who received AI-designed passive plates and those who received no presurgical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Mueller, PhD,MHBA, Study Chair — University Hospital, Basel, Switzerland; Prasad Nalabothu, MDS PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- India (2):
  - Saveetha Medical College, Chennai
  - GSR Hospital Hyderabad, Hyderabad

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications will be shared, including cleft width measurements at birth and at surgery, group assignment, and relevant demographic and clinical variables. A data dictionary defining each variable will be provided. Data will be made available after publication of the primary results upon reasonable request to the study sponsor or principal investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Individual participant data will be made available beginning 6 months after publication of the primary study results and will remain available for a minimum of 3 years following that date. Requests for access can be submitted to the study team during this period.
Access Criteria: Qualified researchers may request access to the de-identified individual participant data for the purpose of academic, non-commercial analyses related to cleft care, digital workflows, or AI-based interventions. Interested investigators must submit a written proposal detailing the research objectives and planned statistical analyses. Requests will be reviewed by the study's data access committee for scientific merit and ethical compliance. Approved researchers will be required to sign a data sharing agreement. Requests can be submitted via email to the principal investigator or designated institutional contact.

REFERENCES:
- [Background] Krozowski ZS, Murphy LC. Stabilisation of the cytoplasmic oestrogen receptor by molybdate. J Steroid Biochem. 1981 Apr;14(4):363-6. doi: 10.1016/0022-4731(81)90155-2. No abstract available. PMID 7230798
- [Background] Benitez BK, Brudnicki A, Surowiec Z, Wieprzowski L, Rasadurai A, Nalabothu P, Lill Y, Mueller AA. Digital impressions from newborns to preschoolers with cleft lip and palate: A two-centers experience. J Plast Reconstr Aesthet Surg. 2022 Nov;75(11):4233-4242. doi: 10.1016/j.bjps.2022.08.015. Epub 2022 Aug 22. PMID 36154982
- [Background] Capizzi SA, Levy NT, Enriquez-Sarano M. Rheumatic fever revisited. Keep this diagnosis on your list of suspects. Postgrad Med. 1997 Dec;102(6):65-6, 71. doi: 10.3810/pgm.1997.12.383. PMID 9406563
- [Background] Meyer S, Benitez BK, Thieringer FM, Mueller AA. Three-Dimensional Printable Open-Source Cleft Lip and Palate Impression Trays: A Single-Impression Workflow. Plast Reconstr Surg. 2024 Feb 1;153(2):462-465. doi: 10.1097/PRS.0000000000010684. Epub 2023 May 15. PMID 37184464
- [Background] Rothman E. Biotechnology overview: where the industry is heading. Healthspan. 1987 Oct;4(9):19-24. No abstract available. PMID 10284965